CLINICAL TRIAL: NCT04397757
Title: An Open-Label, Controlled, Phase 1, Safety and Exploratory Efficacy Study of Convalescent Plasma for Severely Ill, Hospitalized Participants With COVID-19 Pneumonia Caused by SARS-CoV-2.
Brief Title: COVID-19 Convalescent Plasma for the Treatment of Hospitalized Patients With Pneumonia Caused by SARS-CoV-2.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 843003 (PennCCP-02)
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Convalescent plasma
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive either convalescent plasma on Study Day 1 in addition to standard care or standard care alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVID-19 Convalescent plasma (Experimental): COVID-19 Convalescent plasma on Study Day 1 in addition to standard care
  Interventions: Biological: COVID-19 Convalescent Plasma
- Standard care (No Intervention): Standard care alone

INTERVENTIONS:
Biological: COVID-19 Convalescent Plasma — 2 units of COVID-19 convalescent plasma compatible with their blood type
  Arms: COVID-19 Convalescent plasma

SUMMARY:
The purpose of this study is to see if this plasma can be safely used in humans with COVID-19 and to see if it improves patients' health as compared to not using it in patients with pneumonia caused by SARS-CoV-2.

DETAILED DESCRIPTION:
This open-label, randomized, controlled, phase 1 trial will assess the safety and efficacy of convalescent plasma in severely ill, hospitalized participants with pneumonia due to COVID-19. This study will enroll adults 18 years old and older, including pregnant women.

A total of 80 eligible participants will be randomized to receive either 2 units of convalescent plasma collected from ABO-compatible donors who have recovered from COVID-19 and standard of care (treatment arm) or standard of care alone (control arm). Participants in the treatment arm will receive 2 units of convalescent plasma on Study Day 1 in addition to standard of care.

Participants will be assessed on study Day 1 (pre-dose), 30 minutes after each unit of plasma, on all Study Days while hospitalized, and Study Days 15, 22, 29, and 60. All participants will undergo a series of safety and efficacy, assessments. Blood samples will be collected on Days 1 (prior to plasma administration), 3, 8, 15, 29, and 60. Oropharyngeal or endotracheal samples will be collected on Days 1 (prior to plasma administration), 3, 5, 8, 11, and 15.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age
2. Laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other authorized or approved assay in any specimen collected within 72 hours prior to enrollment.

   Note - An exception must be requested to the Sponsor if ≥72 hours since positive test.
3. Hospitalized in participating facility.
4. Documentation of pneumonia with radiographic evidence of infiltrates by imaging (e.g., chest x-ray or CT scan).
5. Abnormal respiratory status that is judged worse than baseline by the investigator and as documented at any point within 24 hours prior to randomization, consistent with ordinal scale levels 5, 6 or 7, specifically defined as:

   * Room air saturation of oxygen (SaO2) < 93%, OR
   * Requiring supplemental oxygen, OR
   * Tachypnea with respiratory rate ≥30
6. Patient or proxy is willing and able to provide written informed consent and comply with all protocol requirements

Exclusion Criteria:

1. Contraindication to transfusion (e.g., severe volume overload, history of severe allergic reaction to blood products), as judged by the investigator.
2. Clinical suspicion that the etiology of acute illness (acute decompensation) is primarily due to a condition other than COVID-19
3. Receipt of other investigational therapy as a part of another clinical trial. Note: investigational therapies used as part of clinical care, (eg, remdesivir, hydroxychloroquine) are permissible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine J. Bar, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Herman JD, Wang C, Burke JS, Zur Y, Compere H, Kang J, Macvicar R, Taylor S, Shin S, Frank I, Siegel D, Tebas P, Choi GH, Shaw PA, Yoon H, Pirofski LA, Julg BD, Bar KJ, Lauffenburger D, Alter G. Nucleocapsid-specific antibody function is associated with therapeutic benefits from COVID-19 convalescent plasma therapy. Cell Rep Med. 2022 Nov 15;3(11):100811. doi: 10.1016/j.xcrm.2022.100811. Epub 2022 Oct 24. PMID 36351430
- [Derived] Bar KJ, Shaw PA, Choi GH, Aqui N, Fesnak A, Yang JB, Soto-Calderon H, Grajales L, Starr J, Andronov M, Mastellone M, Amonu C, Feret G, DeMarshall M, Buchanan M, Caturla M, Gordon J, Wanicur A, Monroy MA, Mampe F, Lindemuth E, Gouma S, Mullin AM, Barilla H, Pronina A, Irwin L, Thomas R, Eichinger RA, Demuth F, Luning Prak ET, Pascual JL, Short WR, Elovitz MA, Baron J, Meyer NJ, Degnan KO, Frank I, Hensley SE, Siegel DL, Tebas P. A randomized controlled study of convalescent plasma for individuals hospitalized with COVID-19 pneumonia. J Clin Invest. 2021 Dec 15;131(24):e155114. doi: 10.1172/JCI155114. PMID 34788233

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-19 Convalescent Plasma: On Day 1 subjects receive 2 units of convalescent plasma collected from ABO-compatible donors who have recovered from COVID-19 followed by standard of care
- Standard of Care: Standard of care treatment administered only
Period: Overall Study
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Started | 41 | 39
Treated | 39 | 39
Completed | 32 | 25
Not Completed | 9 | 14
Not completed — Death | 3 | 11
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Population: One subject (Subject CCP2-043) in treatment plasma arm discontinued/withdrew from study immediately after enrollment before receipt of plasma and was excluded from analysis.
Groups:
- Standard of Care: Standard care alone
- Total: Total of all reporting groups
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 40
  >=65 years | 21 | 18 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 21 | 15 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 21 | 42
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 80

OUTCOME MEASURES:

1. Primary Outcome: Participants With Serious Adverse Events.
Description: Number of participants with at least one serious adverse events (SAEs) up to Study Day 29.
Time Frame: Up to Study Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
Participants | 12 | 15

2. Primary Outcome: Clinical Severity Score
Description: Clinical Severity Score (CSC) measured by both survival time, time to recovery (defined by reaching levels 1-3 of the WHO modified 8-Point Ordinal Severity scale), and disease course while hospitalized and is calculated based on a procedure proposed by Shaw and Fay 2016 (https://doi.org/10.1002/sim.6950). CSC ranges from 1 to 57. Higher CSC is worse outcome.
  Clinical status assessment (WHO modified 8-Point Ordinal Severity scale) includes:
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities and/or requiring home oxygen;
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  5. Hospitalized, requiring supplemental oxygen;
  6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  7. Hospitalized, on invasive mechanical ventilation or ECMO;
  8. Death
Time Frame: Up to Study Day 29
Measure: Median (Inter-Quartile Range); unit: scored on a scale (CSC)
Groups:
- Treatment: On Day 1 subjects receive 2 units of convalescent plasma collected from ABO-compatible donors who have recovered from COVID-19 followed by standard of care
- Control: Standard of care treatment administered only
Arm/Group | Treatment | Control
Number analyzed (Participants) | 40 | 39
scored on a scale (CSC) | 7 [2.75 to 12.5] | 10 [5.5 to 30]

3. Secondary Outcome: Clinical Status Assessment, Time to Recovery
Description: Time to recovery, defined by time needed to reach levels 1-3 using the WHO modified 8-Point Ordinal Severity scale assessed daily while hospitalized and on Day 15, 22, and 29:
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities and/or requiring home oxygen;
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  5. Hospitalized, requiring supplemental oxygen;
  6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  7. Hospitalized, on invasive mechanical ventilation or ECMO;
  8. Death
Time Frame: Up to Study Day 29
Population: Population analyzed are only those who recovered. Remaining subjects either died or were still in hospital with WHO8 score > 3 by Study Day 29.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | COVID-19 Convalescent Plasma | Standard Care
Number analyzed (Participants) | 38 | 26
days | 7 [2.25 to 11.75] | 7 [4.25 to 9.75]

4. Secondary Outcome: National Early Warning Score (NEWS) Clinical Status Assessment
Description: Time to discharge or to a National Early Warning Score (NEWS) of ≤ 2 and maintained for 24 hours, whichever occurs first. NEWS assessed daily while hospitalized until discharge or death and on Days 15 and 29.
  Higher NEWS is worse, range from 0 to 20.
Time Frame: Up to Study Day 29
Population: subjects who never reach National Early Warning Score (NEWS) of ≤ 2 or discharged by Study Day 29 have outcome measure of Infinity
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | COVID-19 Convalescent Plasma | Standard Care
Number analyzed (Participants) | 40 | 39
days | 3 [2 to 6.25] | 4 [2 to 9]

5. Secondary Outcome: Oxygenation
Description: Days of supplemental oxygen while in hospital. defined as days with WHO8 ordinal score of 5, 6, or 7
Time Frame: Daily while hospitalized and up to Study Day 29
Population: All subjects were evaluated. Subjects who never had a day with WHO8 ordinal score of 5, 6, or 7 have outcome measurement of 0 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
days | 7 [2 to 10.25] | 8 [4 to 18.5]

6. Secondary Outcome: Incidence of New Oxygenation Use up to Day 29
Description: Incidence of new oxygenation use up to Day 29.
Time Frame: From enrollment to Day 29.
Population: this endpoint was not measured due to redundancy
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of New Oxygen Use up to Day 29
Description: Duration (days) of new oxygen use up to Day 29.
Time Frame: From enrollment to Day 29.
Population: This was not measured due to redundancy of endpoints
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Non-invasive Ventilation/High Flow Oxygen Days up to Day 29
Description: Days of non-invasive ventilation/high flow oxygen up to Day 29 Defined by having a WHO8 ordinal scale of 6 = Hospitalized, on non-invasive ventilation or high flow oxygen devices
Time Frame: Daily while in hospital to Study Day 29.
Population: All subjects were evaluated. Subjects who never had a day with WHO8 ordinal score of 6 have outcome measurement of 0 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | COVID-19 Convalescent Plasma | Standard Care
Number analyzed (Participants) | 40 | 39
days | 2 [0 to 5] | 3 [0 to 5.5]

9. Secondary Outcome: Number of Participants With at Least One Day on Non-invasive Ventilation/High Flow Oxygen up to Day 29
Description: number of participants with at least one day on non-invasive ventilation/high flow oxygen Defined by having a WHO8 ordinal scale of 6 = Hospitalized, on non-invasive ventilation or high flow oxygen devices
Time Frame: Daily while in hospital until Study Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
Participants | 24 | 23

10. Secondary Outcome: Duration of Non-invasive Ventilation/High Flow Oxygen up to Day 29
Description: Days of non-invasive ventilation/high flow oxygen up to Day 29
Time Frame: Daily while in hospital to Study Day 29.
Population: not measured due to redundancy with other endpoints (#8)
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Ventilator/ECMO Days to Day 29
Description: Days of mechanical ventilation or ECMO use (having a WHO8 ordinal score of 7 = Hospitalized, on invasive mechanical ventilation or ECMO) during the study in hospital until study day 29.
Time Frame: Daily while in hospital to Study Day 29
Population: All subjects were evaluated. Subjects who never had a day with WHO8 ordinal score of 7 have outcome measurement of 0 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
days | 0 [0 to 0] | 0 [0 to 0.5]

12. Secondary Outcome: New Mechanical Ventilation or ECMO Use
Description: number of subjects with new mechanical ventilation or ECMO use up to Day 29 since all subjects were not on mechanical ventilation or ECMO at baseline.
Time Frame: From enrollment to Day 29.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
Participants | 5 | 10

13. Secondary Outcome: Duration of New Mechanical Ventilation or ECMO
Description: Days of new mechanical ventilation or ECMO use up to Day 29.
Time Frame: Daily while in hospital to Study Day 29
Population: only includes subjects with new mechanical ventilation or ECMO
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 5 | 10
days | 7 [4 to 8] | 12.5 [10 to 20.5]

14. Secondary Outcome: Duration of Hospitalization
Description: Duration (days) of first hospitalization. Time until death or discharge or Study Day 29
Time Frame: To Study Day 29
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
days | 7 [2.75 to 12] | 9 [5 to 19.5]

15. Secondary Outcome: Mortality
Description: 28 day mortality.
Time Frame: 28 days from Study Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
Participants | 2 | 10

16. Secondary Outcome: Number of Subjects With SAEs Through Day 29
Description: Number of subjects with SAEs through Day 29.
Time Frame: Through Study Day 29
Population: this endpoint is redundant with the primary endpoint
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Subjects With at Least One Grade 3 and Grade 4 Clinical and/or Laboratory Adverse Events Through Day 29
Description: Number of subjects with at least one Grade 3 or Grade 4 clinical and/or laboratory adverse events (AEs) through Day 29.
Time Frame: Through Study Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
Participants | 18 | 22

18. Secondary Outcome: Changes in WBC With Differential Through Day 29
Description: Collected labs on Days 1 (baseline), 3, 5, 8, and 11 (while hospitalized), Days 15 and 29 (if attends in person visit or still hospitalized). Changes measured as difference between last measured lab value and baseline lab value. A negative value indicates last lab value > baseline lab value.
Time Frame: Through Day 29
Population: Defined changes as difference between last measured lab value and baseline (day 1) lab value. Day of last measured lab may differ among subjects.
Measure: Median (Inter-Quartile Range); unit: THO/uL
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
THO/uL | 1.45 [-1.30 to 3.30] | 2.50 [0.25 to 3.30]

19. Secondary Outcome: Changes in Hemoglobin Measurement Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
g/dL | -0.35 [-1.20 to 0.325] | -0.30 [-1.90 to 0.90]

20. Secondary Outcome: Changes in Platelets Measurement Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: 10^3 platelets per uL
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
10^3 platelets per uL | 38 [-5.50 to 129] | 59 [4.50 to 94.50]

21. Secondary Outcome: Changes in Creatinine Measurement Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
mg/dL | 0.035 [-0.160 to 0.220] | -0.050 [-0.255 to 0.055]

22. Secondary Outcome: Changes in Glucose Measurement Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 39
mg/dL | -14.00 [-34.75 to 13.75] | -20.00 [-48.50 to 5.00]

23. Secondary Outcome: Changes in Total Bilirubin Measurement Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29
Population: Defined changes as difference between last measured lab value and baseline (day 1) lab value. Day of last measured lab may differ among subjects.
  Standard of care arm has analyzed sample size of 38 because one subject did not have total bilirubin lab collected
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 38
mg/dL | 0.00 [-0.10 to 0.10] | 0.00 [0.00 to 0.10]

24. Secondary Outcome: Changes in ALT Measurement Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29
Population: Defined changes as difference between last measured lab value and baseline (day 1) lab value. Day of last measured lab may differ among subjects.
  Standard of care arm has analyzed sample size of 38 because one subject did not have ALT lab collected
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 38
U/L | 0.00 [-5.75 to 5.00] | -1.00 [-11.50 to 8.25]

25. Secondary Outcome: Changes in AST Measurement Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29.
Population: Defined changes as difference between last measured lab value and baseline (day 1) lab value. Day of last measured lab may differ among subjects.
  Standard of care arm has analyzed sample size of 38 because one subject did not have AST lab collected
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 40 | 38
U/L | -7.00 [-16.00 to 0.00] | -6.00 [-16.00 to 0.75]

26. Secondary Outcome: Changes in PT Measurement Laboratory Through Day 29
Description: as for outcome 18
Time Frame: Through Day 29.
Population: Defined changes as difference between last measured lab value and baseline (day 1) lab value. Day of last measured lab may differ among subjects.
  Plasma arm analyzed sample size is 38 because 2 subjects did not have PT test collected.
  Standard of care arm analyzed sample size is 37 because 2 subjects did not have PT test collected.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | COVID-19 Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 38 | 37
seconds | 0.0 [-1.175 to 0.550] | 0.0 [-0.8 to 1.2]

ADVERSE EVENTS:
Time Frame: Up to Study Day 60
Description: 41 subjects were enrolled in the treatment arm; 1 subject withdrew consent prior to initiate any research activities; Only 40 were placed at risk.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 3/40 | 11/39
Serious Adverse Events (participants affected / at risk) | 13/40 | 19/39
Other Adverse Events (participants affected / at risk) | 15/40 | 20/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (N=40) | Control (N=39)
Acute CNS Ischemia (Vascular disorders) | 2 (2) | 1 (1) — Transient ischemic attack; cerebral vascular accident
Altered Mental Status (Nervous system disorders) | 1 (1) | 1 (1)
Arrhythmia (by ECG or physical examination) (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine High (Investigations) | 0 (0) | 1 (1) — Creatinine greater than 2x baseline
Glucose low (Endocrine disorders) | 0 (0) | 1/32 (1)
Dyspnea or Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 13 (18)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (3)
Pain (General disorders) | 3 (3) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neurosensory alteration (Nervous system disorders) | 0 (0) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=40) | Control (N=39)
Acidosis (Metabolism and nutrition disorders) | 6 (7) | 4 (4)
Albumin, Low (Metabolism and nutrition disorders) | 2 (3) | 4 (4)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Altered Mental Status (Nervous system disorders) | 2 (2) | 5 (5)
Arrhythmia (by ECG or physical examination) (Cardiac disorders) | 0 (0) | 5 (5)
AST, High (Investigations) | 2 (2) | 2 (2)
Blood Pressure Abnormalities Hypertension (with the lowest reading taken after repeat testing durin (Vascular disorders) | 1 (1) | 8 (11)
Creatinine, High (Investigations) | 4 (4) | 5 (6)
Dyspnea or Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 14 (32)
Fever (non-axillary temperatures only) (General disorders) | 3 (4) | 5 (7)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2)
Glucose (mg/dL; mmol/L) Fasting, High (Metabolism and nutrition disorders) | 5 (6) | 7 (9)
Hematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Hemoglobin, Low (g/dL; mmol/L) >= 13 years of age (female only) (Blood and lymphatic system disorders) | 6 (9) | 8 (14)
Hypotension (Vascular disorders) | 4 (4) | 7 (9)
Platelets, Decreased (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Acute CNS Ischemia (Nervous system disorders) | 1 (1) | 2 (3)
ALT High (Investigations) | 0 (0) | 2 (2)
Calcium, Low (mg/dL; mmol/L) >= 7 days of age (Investigations) | 1 (1) | 2 (2)
Hemoglobin, Low (g/dL; mmol/L) >= 13 years of age (male only) (Blood and lymphatic system disorders) | 4 (4) | 6 (10)
Pain (not associated with study agent injections and not specified elsewhere) (General disorders) | 1 (1) | 2 (2)
Pruritus (without skin lesions) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Thrombosis or Embolism Report only one (Blood and lymphatic system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT04397757/Prot_SAP_000.pdf